CLINICAL TRIAL: NCT04919512
Title: A Phase 2, Open-Label, Multi-Center, Randomized Study of TAR-200 in Combination With Cetrelimab and Cetrelimab Alone in Participants With Muscle-Invasive Urothelial Carcinoma of the Bladder Who Are Scheduled for Radical Cystectomy and Are Ineligible for or Refusing Platinum-Based Neoadjuvant Chemotherapy
Brief Title: A Study of TAR-200 in Combination With Cetrelimab and Cetrelimab Alone in Participants With Muscle-Invasive Urothelial Carcinoma of the Bladder
Acronym: SunRISe-4
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109044; 17000139BLC2002 (Other: Janssen Research & Development, LLC); 2020-005565-13 (EudraCT Number)
Expanded Access: NCT06877676 (Approved for marketing)
Record Dates: First submitted 2021-06-08; First posted 2021-06-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: TAR-200 + Cetrelimab (Experimental): Participants will receive TAR-200 in combination with cetrelimab.
  Interventions: Drug: TAR-200; Biological: Cetrelimab
- Cohort 2: Cetrelimab (Experimental): Participants will receive cetrelimab.
  Interventions: Biological: Cetrelimab

INTERVENTIONS:
Drug: TAR-200 — TAR-200 will be administered.
  Other Names: JNJ-17000139
  Arms: Cohort 1: TAR-200 + Cetrelimab
Biological: Cetrelimab — Cetrelimab will be administered.
  Other Names: JNJ-63723283

SUMMARY:
The purpose of this study is to evaluate the anti-tumor effects of TAR-200 in combination with intravenous (IV) cetrelimab and IV cetrelimab alone.

DETAILED DESCRIPTION:
Bladder cancer is the tenth most common malignancy worldwide. Approximately 25 percent (%) of all new bladder cancer participants present with muscle invasive bladder cancer (MIBC) at the time of diagnosis, and roughly 50% will ultimately develop distant metastases. The TAR-200/ gemcitabine (JNJ-17000139) product is an intravesical drug delivery system regulated as an investigational drug. The drug constituent consists of gemcitabine minitablets and osmotic minitablets. Cetrelimab (JNJ-63723283) is a fully human immunoglobulin G4 (IgG4) kappa monoclonal antibody (mAb) that binds programmed-cell death protein (PD)-1. The standard of care in MIBC includes radical cystectomy (RC) with urinary diversion and is considered the preferred treatment option for participants who are considered surgical candidates. Study consists of a Screening phase, Treatment phase and follow-up phase. The total duration of study will be up to 2 years and 6 months. Efficacy, safety, pharmacokinetics (PK), and biomarkers will be assessed at specific time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, cT2-T4a N0, M0 infiltrating urothelial carcinoma of the bladder. Initial diagnosis must have been within 120 days of randomization date. Participants with variant histologic subtypes are allowed if tumor(s) demonstrate urothelial predominance. However, the presence of small cell or neuroendocrine variants will make a participant ineligible
* Participants with no residual tumor, or intravesical tumor size of less than or equal to (<=)3 centimeter (cm) following transurethral resection of bladder tumor (TURBT) are eligible; debulking TURBT for any residual disease is encouraged but not mandated. Participants with persistent tumors greater than (>)3 cm at screening must undergo a second debulking, re-staging TURBT. Participants will be ineligible if any individual tumor is >3 cm after debulking TURBT
* Deemed eligible for and willing to undergo RC by the operating urologist
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0 or 1
* Thyroid function tests within normal range or stable on hormone supplementation per investigator assessment. Investigators may consult an endocrinologist for participant eligibility assessment in the case of equivocal or marginal tests results
* All adverse events associated with any prior surgery must have resolved to common terminology criteria for adverse events (CTCAE) version 5.0 Grade less than (<) 2 prior to randomization

Exclusion Criteria:

* Must not have received prior systemic chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to starting study treatment
* Participants must not have evidence of cT4b, or N1-3, or M1 disease based on central radiology staging (chest, abdomen, and pelvis must be performed using computed tomography [CT] or magnetic resonance imaging [MRI]) within 42 days prior to randomization
* Presence of any bladder or urethral anatomic feature that, in the opinion of the Investigator, may prevent the safe placement, indwelling use, or removal of TAR-200
* Prior systemic chemotherapy for urothelial cell carcinoma of the bladder at any time
* Currently participating or has participated in a study of an investigational agent and received study therapy or investigational device within 4 weeks prior to enrollment
* Participants with evidence of bladder perforation during diagnostic cystoscopy. Participant is eligible if perforation has resolved prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Pathologic Complete Response (pCR) | Up to Week 15
  Percentage of participants with a pathologic complete response (pCR) or no evidence of pathologic intravesical disease and nodal involvement (ypT0N0) derived from analysis of radical cystectomy (RC) bladder specimen will be reported.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to Week 108
  RFS is defined as the time from first dose of any study treatment to first radiologic (as assessed by response evaluation criteria in solid tumors [RECIST] 1.1 criteria) or histologic evidence of nodal or metastatic disease or death due to any cause.
Number of Participants with Adverse Events (AEs) by Grades According to Common Terminology Criteria for Adverse Events (CTCAE) | Up to Week 108
  Number of participants with AEs by severity grade as assessed by CTCAE version 5 will be reported. Grade refers to the severity of AE as follows: Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5- Death related to adverse event.
Number of Participants with Change from Baseline in Laboratory Abnormalities | Up to Week 108
  Number of participants with change from baseline in laboratory abnormalities will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (109):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - UAMS Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - Arkansas Urology, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Genesis Research, San Diego, California
  - Colorodo Urology- St. Anthony Hospital, Golden, Colorado
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - DuPage Medical Group, Lisle, Illinois
  - Urology of Indiana, Indianapolis, Indiana
  - First Urology, Jeffersonville, Indiana
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Penn Medicine - PerelmanCenter for Advanced Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Institute of Urology, PC, Troy, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University School Of Medicine - Center For Advanced Medicine (CAM), St Louis, Missouri
  - David C. Pratt Cancer Center, St Louis, Missouri
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Mount Sinai Queens Infusion Center, Astoria, New York
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Associated Medical Professionals, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington School of Medicine, Seattle, Washington
- Belgium (6):
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Hopital de Jolimont, Haine Saint Paul La Louviere
  - ZNA Jan Palfijn, Merksem
  - Centre Interuniversitaire Ambroise Pare - Ambroise Paré, Mons
- France (14):
  - Clinique Tivoli Ducos, Bordeaux
  - ICH Hopital A. Morvan, Brest
  - Hopital Henri Mondor, Créteil
  - Hôpital Privé Le Bois, Lille
  - Polyclinique de Limoges - Francois Chenieux, Limoges
  - Hopital de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - Hopital Europeen Georges-Pompidou, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - Clinical La Croix Du Sud - Ramsay Santé, Quint-Fonsegrives
  - HIA se Sainte-Anne - Toulon, Toulon
  - Clinique Pasteur, Toulouse
- Germany (6):
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt am Main
  - Universitaetsklinikum Halle Saale, Halle
  - Marien hospital Herne, Herne
  - Vivantes Klinikum Am Urban, Kreuzberg
  - Universitatsklinikum Munster, Münster
- Israel (6):
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center - Hasharon Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Ospedale San Giuseppe Moscati di Avellino, Avellino
  - Ospedale Civile Ramazzini, Carpi
  - SPDC Villa Scassi, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Dei Tumori Di Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - ASL Napoli 2 Nord-SM delle Grazie Hospital, Pozzuoli
  - Istituto Nazionale Tumori Regina Elena, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Netherlands (4):
  - Ziekenhuisgroep Twente, Almelo
  - Radboud Umcn, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Haga ziekenhuis, The Hague
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Samsung Medical Center, Gangnam Gu
  - National Cancer Center, Goyang-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (7):
  - Hosp Univ A Coruna, A Coruña
  - Fund. Puigvert, Barcelona
  - Hosp. Univ. San Cecilio, Granada
  - Clinica Univ. de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Lancashire Teaching Hospitals NHS Foundation Trust Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Necchi A, Guerrero-Ramos F, Crispen PL, Herrera-Imbroda B, Garje R, Szabados B, Peyton CC, Pradere B, Ku JH, Shore N, Bogemann M, Preston MA, Xylinas E, Sanchez de Llano C, Gong C, Hasan M, Urtishak K, Battaglia S, Stitou H, Bhanvadia S, Sweiti H, Psutka SP. Gemcitabine Intravesical System Plus Cetrelimab or Cetrelimab Alone as Neoadjuvant Therapy in Muscle-Invasive Bladder Cancer: SunRISe-4 Primary Analysis and Biomarker Results. J Clin Oncol. 2025 Dec 3:JCO2502382. doi: 10.1200/JCO-25-02382. Online ahead of print. PMID 41337691
- [Derived] Necchi A, Guerrero-Ramos F, Crispen PL, Herrera-Imbroda B, Garje R, Powles T, Peyton CC, Pradere B, Ku JH, Shore N, Bogemann M, Preston MA, Xylinas E, Sanchez de Llano C, Hasan M, Stitou H, Bhanvadia S, Sweiti H, Psutka SP. TAR-200 plus cetrelimab versus cetrelimab monotherapy as neoadjuvant therapy in patients with muscle-invasive bladder cancer who are ineligible for or decline neoadjuvant cisplatin-based chemotherapy (SunRISe-4): interim analysis of a randomised, open-label phase 2 trial. Lancet Oncol. 2025 Oct;26(10):1312-1322. doi: 10.1016/S1470-2045(25)00358-4. Epub 2025 Aug 27. PMID 40885199